CLINICAL TRIAL: NCT06309303
Title: Clinical Features and Manifestations of Kawasaki Disease During the SARS-COV-2 Epidemic
Brief Title: Kawasaki Disease During the COVID-19 Epidemic
Acronym: KAWACOVID
Status: Completed | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 12/20
Record Dates: First submitted 2023-03-29; First posted 2024-03-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Kawasaki Disease
Keywords: Kawasaki Disease; SARS-COV-2; Children
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- KD with SARS-COV-2: Subjects with Kawasaki Disease and presence of concomitant SARS-COV-2 infection
  Interventions: Other: Clinical evaluation
- KD without SARS-COV-2: Subjects with Kawasaki Disease and absence of concomitant SARS-COV-2 infection
  Interventions: Other: Clinical evaluation

INTERVENTIONS:
Other: Clinical evaluation — Evaluation of clinical manifestation, laboratory ad imaging testing results, disease course, treatment and outcome

SUMMARY:
Northern Italy is the second region hit by the SARS-COV2 infection worldwide. Data on COVID-19 clinical presentation in children is still scarce, but fewer rate of infection and milder disease seem typical of this age group. In the last three weeks it has been reported an abnormal number of critically ill patients with clinical characteristics consistent with Kawasaki Shock Syndrome (KSS). The common manifestations are: "middle aged" children (6-9 y/o) with a history of persistent high spiking fever in the last days, abdominal pain, diarrhea, skin rash and rapidly deteriorating clinical condition with the onset of shock, without clear signs of dehydration. Other less common features are arthralgia, cough, meningism, conjunctivitis and reddened, cracked lips. Labworks usually show high inflammatory markers, low lymphocyte counts, low sodium, and high troponin levels. Echocardiography have been consistent with myocarditis in the majority of patient instead of classical coronary artery abnormalities. Patients have been diagnosed as Kawasaki disease (typical or incomplete) and treated accordingly with IntraVenous ImmunoGlobulin (IVIG) and/or steroids. One patient refractory to such treatments responded successfully to intravenous Anakinra. All the patients reported a family history consistent with COVID-19, serology and naso-pharyngeal swabs were inconsistently positive. To date we are aware of at least 10 such cases. KSS is a rare and dreadful complication, with an estimated prevalence of 5% of patients with Kawasaki Disease (KD). Given the extreme rarity of this condition, the occurrence of so many cases in the last weeks points to a possible causative agent. As our hospitals are in high endemic area, SARS-COV2 seems the most obvious, although testing for such infection in patients returned conflicting results. It is not clear, at this moment, if this clinical entity is a proper KD triggered by SARS-COV2, or a systemic vasculitis with similar features of KD, secondary to SARS-COV2 infection. The aim of this nationwide study is to better define this clinical entity.

ELIGIBILITY:
Inclusion Criteria:

* All children with clinical diagnosis of Kawasaki Disease
* age<18 years
* Absence of other underlying chronic diseases

Exclusion Criteria:

* Presence of underlying chronic diseases
* Not fulfilling clinical criteria for Kawasaki Disease diagnosis

Ages: 1 Month to 18 Months | Sex: All
Age Groups: Child
Study Population: Children (age 0-17 years) affected by Kawasaki Disease
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Kawasaki Disease and concomitant SARS-COV-2 infection | Through study completion, an average of 4 months
  Subjects with KD-like multi-inflammatory syndrome diagnosis, named as KawaCOVID Group based on the presence of 1) persistent fever (> 48 h), lymphopenia and evidence of single or multi-organ dysfunction with other additional clinical, laboratory or imagining; 2) exclusion of any other microbial cause will be identified.

SECONDARY OUTCOMES:
Number of subjects with Kawasaki Disease without concomitant SARS-COV-2 infection | Through study completion, an average of 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Taddio, MD, Study Director — IRCCS materno infantile Burlo Garofolo
Locations (4):
- Italy (4):
  - Ospedale Pediatrico Meyer, Florence
  - IRCCS Istituto Giannina Gaslini, Genova
  - Ospedale Pediatrico Bambino Gesù, Roma
  - IRCCS Burlo Garofolo, Trieste

IPD SHARING:
Plan to Share IPD: Undecided